CLINICAL TRIAL: NCT02179931
Title: Interventional, Single Dose, Open-label, Randomised, Crossover, Bioequivalence Study in Healthy Men and Women to Compare Two Pharmaceutical Formulations of Flupentixol/Melitracen (Deanxit®)
Brief Title: Bioequivalence Study in Healthy Men and Women to Compare Two Pharmaceutical Formulations of Flupentixol/Melitracen (Deanxit®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15972A; 2014-000431-17 (EudraCT Number)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Men and Women
MeSH Terms: interventions — Flupenthixol; flupentixol, melitracen drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flupentixol/melitracen film-coated tablet (Experimental): test treatment - 0.5 mg/10 mg; oral as a single dose
  Interventions: Drug: Flupentixol/melitracen film-coated tablet
- Flupentixol/melitracen coated tablet (Deanxit®) (Other): reference treatment - 0.5 mg/10 mg, oral as a single dose
  Interventions: Drug: Flupentixol/melitracen coated tablet (Deanxit®)

INTERVENTIONS:
Drug: Flupentixol/melitracen film-coated tablet
  Arms: Flupentixol/melitracen film-coated tablet
Drug: Flupentixol/melitracen coated tablet (Deanxit®)
  Arms: Flupentixol/melitracen coated tablet (Deanxit®)

SUMMARY:
To establish bioequivalence of flupentixol/melitracen between a new film-coated tablet formulation of 0.5 mg flupentixol/10 mg melitracen and the marketed coated tablet formulation of 0.5 mg flupentixol/10 mg melitracen (Deanxit®), administered as single doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥18 and ≤55 years of age with a body mass index (BMI) of >18.5 and <30 kg/m2.
* Women will be non-pregnant and non-lactating.

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area under the flupentixol plasma concentration-time curve from zero to 72 hours post dose (AUC0-72h) | Up to 72 hours post dose
Maximum observed concentration (Cmax) of flupentixol | Up to 312 hours post dose
Area under the melitracen plasma concentration-time curve from zero to 72 hours post dose (AUC0-72h) | Up to 72 hours post dose
Maximum observed concentration (Cmax) of melitracen | Up to 312 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom